CLINICAL TRIAL: NCT05059743
Title: Single Dose Absorption, Distribution, Metabolism, and Excretion Study of [14C] - Larotinib in Healthy Male Participants
Brief Title: ADME Study of [14C]- Larotinib in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Z650-HV-106
Record Dates: First submitted 2021-09-15; First posted 2021-09-28 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2021-09

CONDITIONS: Healthy Adult Male Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]-Larotinib (Experimental): Patients will receive single dose of [14C]-Larotinib (Suspension, 350mg/100μCi).
  Interventions: Drug: [14C]-Larotinib

INTERVENTIONS:
Drug: [14C]-Larotinib — Patients will receive single dose of orally [14C]-Larotinib on Day 1.

SUMMARY:
Study to Evaluate the Mass Balance and Biotransformation of Single Dose [14C]-Larotinib（Z650）in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males, 18 to 45 years at the time of screening.
* Weight>50 kg, Body mass index (BMI) is 19~26 kg/m2
* signing of informed consent
* Volunteers are able to communicate well with the investigators and be able to complete the trial according to the process

Exclusion Criteria:

* physical examination, vital signs, routine laboratory tests 12-lead ECG, Chest X-ray ,ophthalmologic examination, abdominal B-ultrasound and other abnormalities and clinical significance.
* positive testing for HIV, HBsAg, HBeAb, HCVAb or Syphilis antibody.
* C- reactive protein (CRP) abnormalities are clinically significant or New Coronavirus nucleic acid positive.
* Screening for use of any clinical trial drug within the first 3 months or withdrawal time shorter than the 7 half-life period of the trial drug at enrollment, whichever is the longest of the two;
* CYP3A4, CYP2C8 , CYP2C9 and p-gp inducers or inhibitors were taken within 28 days before screening
* Use of any prescription or over-the-counter drug, any vitamin product, health care drug or Chinese herbal medicine within 14 days prior to screening;
* clinical symptoms or diseases of the heart;supraventral or ventricular arrhythmia with clinical significance that requires treatment or intervention; QTcF>450ms at screening stage
* Patients who had undergone major surgery or whose surgical incision was not completely healed within 6 months before the screening period;Major surgery includes, but is not limited to, any surgery with a significant risk of bleeding, prolonged general anesthesia, or an open biopsy or significant traumatic injury;
* Significant clinical bleeding symptoms or definite bleeding tendency occurred within 3 months before screening
* Screening for abdominal fistula, gastrointestinal perforation or abdominal abscess in the first 6 months;
* Hemorrhoids or perianal diseases with regular/bleeding in the stool;Patients with gastrointestinal dysfunction, such as irritable bowel syndrome and inflammatory bowel disease, may be affected by drug absorption as determined by researchers;
* Allergic persons,
* A history of any clinically serious illness or condition, including but not limited to circulatory, endocrine, nervous, digestive, urinary, or blood, immune, mental, and metabolic diseases, that the investigator considers to be likely to affect the results of the study;
* Habitual constipation or diarrhea;
* Heavy drinking or regular drinking in the six months preceding the screening period
* Those who had smoked more than 5 cigarettes per day on average in the 3 months before the screening period or habitually used nicotine-containing products and were unable to quit during the test period;
* Substance abuse or use of soft drugs (e.g., marijuana) in the 3 months prior to the screening period or use of hard drugs (e.g., cocaine, amphetamines, phenylcyclohexidine, etc.) in the 1 year prior to the screening period;Or screening for positive urine drug abuse (drug) tests;
* habitual consumption of grapefruit juice or excessive consumption of tea, coffee and/or caffeinated beverages and failure to abstain during the study period;
* Those with a history of fainting needle or blood, have difficulty in blood collection or cannot tolerate vein puncture for blood collection;
* Workers engaged in conditions requiring long-term exposure to radioactivity;Or have significant radiation exposure (≥2 chest/abdomen CT, or ≥3 other types of X-ray examinations) within 1 year before the test or have participated in the radiopharmaceutical labeling test;
* Those who have lost blood or donated up to 400 mL within 3 months before the screening period, or those who have received blood transfusion, or those who plan to donate blood within 3 month after the end of this test;
* Those who have been vaccinated within 1 month before screening or those who plan to be vaccinated during the trial period;
* Having family planning during the trial period and within 12 months after the last use of the drug, or not agreeing that subjects and their spouses should take strict contraceptive measures during the trial period and within 12 months after the last use of the drug;
* As determined by the investigator, the subject has other factors that are not suitable for the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2021-11-20 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Cumulative excretion of 14C-labeled drug-related material (radioactivity in plasma, urine and fecal samples) | up to 15 days
  Percent (%) of each radiolabeled drug-related material (parent and each metabolite) will be determined in plasma, urine and feces.
Identification of the Proportion of different metabolites to determine biotransformation pathway of Larotinib | up to 15 days
  Proportion of different metabolites(Larotinib and main metabolites） .

SECONDARY OUTCOMES:
Quantitive analysis of the concentrations of Larotinib in plasma using the validated LC-MS/MS to obtain pharmacokinetic data | up to 15 days
  The concentrations of Larotinib in plasma
Adverse events | up to 22 days
  Adverse events assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: liyan Miao, MD, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China